CLINICAL TRIAL: NCT03810417
Title: Single System Double Blinded Trial to Evaluate the Effect of Pre-operative Treatment With DigiFab to Prevent Post-operative Acute Kidney Injury (AKI) in Patients at High Risk for AKI Undergoing Cardiac Bypass Graft Surgery
Brief Title: Preop Digifab in CABG to Reduce Ouabain Levels and Prevent AKI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Stephen Gottlieb, Professor of Medicine, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HP-00083553
Record Dates: First submitted 2019-01-08; First posted 2019-01-18 (Actual); Results first posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Acute Kidney Injury
Keywords: coronary artery bypass surgery; ouabain; acute kidney injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — digoxin antibodies Fab fragments

STUDY DESIGN:
Intervention Model Description: Patients undergoing coronary artery bypass surgery
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigational pharmacy will provide active drug or placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Digifab, EO > 360 (Active Comparator): Digifab intravenous in subject with baseline ouabain concentration > 360 pm
  Interventions: Drug: Digoxin Antibodies Fab Fragments; Diagnostic Test: Baseline EO > 360 pM
- Placebo, EO > 360 (Placebo Comparator): saline intravenous n subject with baseline ouabain concentration > 360 pm
  Interventions: Other: Placebo; Diagnostic Test: Baseline EO > 360 pM
- Digifab, EO < 360 (Active Comparator): Digifab in subject with baseline ouabain concentration < 360 pm
  Interventions: Drug: Digoxin Antibodies Fab Fragments; Diagnostic Test: EO < 360 pM
- Placebo, EO < 360 (Placebo Comparator): Subjects who received Placebo in n subject with baseline ouabain concentration < 360 pm
  Interventions: Other: Placebo; Diagnostic Test: EO < 360 pM

INTERVENTIONS:
Drug: Digoxin Antibodies Fab Fragments — Digoxin antibodies
  Arms: Digifab, EO < 360; Digifab, EO > 360
Other: Placebo — Saline
  Arms: Placebo, EO < 360; Placebo, EO > 360
Diagnostic Test: Baseline EO > 360 pM — Baseline ouabain concentration > 360 pM
  Arms: Digifab, EO > 360; Placebo, EO > 360
Diagnostic Test: EO < 360 pM — Baseline ouabain concentration < 360 pM
  Arms: Digifab, EO < 360; Placebo, EO < 360

SUMMARY:
Acute kidney injury (AKI) occurs in up to 30% of patients undergoing coronary artery bypass graft (CABG) surgery, and often requires patients to go on dialysis. In patients needing dialysis, the risk of dying is very high.There are no known therapies to reduce the chance of developing kidney damage after heart surgery. There is evidence that patients with high levels of a substance called ouabain have an increased risk of developing kidney damage. This study is testing the hypothesis that giving a medication called DigiFab to lower the ouabain levels will reduce the risk of developing kidney damage after heart surgery.

DETAILED DESCRIPTION:
This is a randomized double-blinded study investigating the role of DigiFab in patients with elevated risk of acute kidney injury undergoing CABG surgery. University of Maryland Medical Center (UMMC) and University of Maryland St Joseph Medical Center (UMSJMC) patients who are undergoing CABG, meet the inclusion criteria and provide consent will be enrolled in this study and randomized to either DigiFab arm or the placebo (vehicle) arm. The study involves a follow up period of 72 hours post CABG surgery.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing coronary artery bypass surgery
* glomerular filtration rate > 15 History of Diabetes Mellitus or GFR < 60

Exclusion Criteria:

* Allergy to Digifab Contrast dye within 3 days Creatinine > 25% above baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen S Gottlieb, Principal Investigator — University of Maryland
Locations (2):
- United States (2):
  - University of Maryland, Baltimore, Maryland
  - St Josephs Medical Center, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients randomized and double blinded
Groups:
- Digifab Below Median: Received Digifab with baseline ouabain below 360 pm
- Placebo Below Median: Received placebo with baseline ouabain below 360 pm
- Digifab Above Median: Digifab intravenous with baseline ouabain above 360 pm
- Placebo Above Median: saline intravenous with baseline ouabain above 360 pm
Period: Overall Study
Arm/Group | Digifab Below Median | Placebo Below Median | Digifab Above Median | Placebo Above Median
Started | 70 | 64 | 64 | 69
Completed | 66 | 59 | 59 | 66
Not Completed | 4 | 5 | 5 | 3

BASELINE CHARACTERISTICS:
Population: As per the protocol, The only patients analyzed are those who received study drug,and had surgery. Therefore 250 patients were analyzed
Groups:
- Digifab Below Median: Received Digifab with baseline ouabain below median
- Placebo Below Median: Received placebo with baseline ouabain below median
- Digifab Above Median: Digifab intravenous with baseline ouabain above median
- Placebo Above Median: saline intravenous with baseline ouabain above median
- Total: Total of all reporting groups
Arm/Group | Digifab Below Median | Placebo Below Median | Digifab Above Median | Placebo Above Median | Total
Number analyzed (Participants) | 70 | 64 | 64 | 69 | 267
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Agre (years) Population: Only patients who received study drug and had surgery were analyzed. 17 patients randomized did not fulfil these requirements
  years
    number analyzed (Participants) | 66 | 59 | 59 | 66 | 250
    (all) | 66 [60 to 71] | 67 [63 to 74] | 65 [59 to 74] | 70 [62 to 74] | 67 [61 to 73]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Only patients who received study drug and had surgery were analyzed, as per the protocol.
  Participants
    number analyzed (Participants) | 66 | 59 | 59 | 66 | 250
    Female | 15 | 14 | 15 | 16 | 60
    Male | 51 | 45 | 44 | 50 | 190
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Only patients who received study drug and had surgery were analyzed, as per the protocol.
  Participants
    number analyzed (Participants) | 66 | 59 | 59 | 66 | 250
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Asian | 1 | 4 | 1 | 2 | 8
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 9 | 16 | 9 | 5 | 39
    White | 54 | 39 | 49 | 59 | 201
    More than one race | 1 | 0 | 0 | 0 | 1
    Unknown or Not Reported | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Renal Function
Description: Change in glomerular filtration rate (measured by Cockcroft-Gault Formula), mL/min per 1.73 m2 from baseline to 72 hours
Time Frame: 72 hours
Population: Randomized study with endpoint assessed in those with baseline ouabain concentration (EO) above and below 360 pM
Measure: Median (Inter-Quartile Range); unit: mL/min/1.73m^2
Groups:
- Digifab, EO > 360: Received Digifab and had a baseline EO concentration > 360
- Placebo, EO > 360: Received placebo and had a baseline EO concentration > 360
- Digifab, Eo < 360: Subjects who received digifab and had baseline ouabain < 360
- Placebo, EO < 360: Subjects who received placebo and had a baseline ouabain < 360
Arm/Group | Digifab, EO > 360 | Placebo, EO > 360 | Digifab, Eo < 360 | Placebo, EO < 360
Number analyzed (Participants) | 59 | 66 | 66 | 59
mL/min/1.73m^2 | .46 [-7.4 to 7.5] | .75 [-9.1 to 6.2] | 4.26 [-0.89 to 11.59] | 2.80 [-4.07 to 13.17]
Statistical Analysis 1: Comparison: Digifab, EO > 360 vs Placebo, EO > 360; Test type: Superiority; p > 0.05, Regression, Linear
Statistical Analysis 2: Comparison: Digifab, EO > 360 vs Placebo, EO > 360; Test type: Superiority; p < 0.05, Regression, Logistic

2. Secondary Outcome: AKI
Description: Development of AKI at 72 hours
Time Frame: 3 days
Population: Results by intervention and baseline ouabain concentration
Measure: Number; unit: participants
Groups:
- Digifab > 360: Subjects who received digifab and had baseline ouabain > 360
- Placebo > 360: Subjects who received placebo and had baseline ouabain > 360
- Digifab < 360: Subjects who received digifab and had baseline ouabain < 360
- Placebo < 360: Subjects who received placebo and had baseline ouabain < 360
Arm/Group | Digifab > 360 | Placebo > 360 | Digifab < 360 | Placebo < 360
Number analyzed (Participants) | 59 | 66 | 66 | 59
participants | 5 | 12 | 8 | 8

ADVERSE EVENTS:
Time Frame: 30 days
Groups:
- Digifab and EO > 360 pM: Received Digifab and baseline ouabain concentration > 360 pM
- Placebo, EO > 360 p: Received placebo and baseline ouabain concentration > 360 pM
- Digifab and EO < 360 pM: Received Digifab and baseline ouabain concentration < 360 pM
- Placebo, EO < 360 pM: Received placebo and baseline ouabain concentration< 360 pM
Arm/Group | Digifab and EO > 360 pM | Placebo, EO > 360 p | Digifab and EO < 360 pM | Placebo, EO < 360 pM
All-Cause Mortality (participants affected / at risk) | 0/59 | 2/66 | 1/66 | 2/59
Serious Adverse Events (participants affected / at risk) | 17/59 | 20/66 | 14/66 | 16/59
Other Adverse Events (participants affected / at risk) | 0/59 | 0/66 | 0/66 | 0/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Digifab and EO > 360 pM (N=59) | Placebo, EO > 360 p (N=66) | Digifab and EO < 360 pM (N=66) | Placebo, EO < 360 pM (N=59)
Diverse (Cardiac disorders) | 17 (30) | 20 (39) | 14 (27) | 16 (31) — Secondary to surgery

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-24): https://cdn.clinicaltrials.gov/large-docs/17/NCT03810417/Prot_SAP_001.pdf